CLINICAL TRIAL: NCT02991534
Title: Facilitating Cardiovascular Risk Screening and Risk Reduction in Women Veterans (QUE 15-272)
Brief Title: Cardiovascular Risk Screening and Risk Reduction in Women Vets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 16-007
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases; Hypertension; Hyperlipidemias; Dyslipidemias; Obesity; Diabetes Mellitus; Tobacco Use Disorder; Overweight
Keywords: Patient Participation [N05.300.150.600.620]; Health Behavior [F01.145.488]; Women [M01.975]; Patient Satisfaction [N05.715.360.600]; Physicians, Primary Care [M01.526.485.810.800]; Physicians, Women [M01.526.485.810.820]; Health Educators [M01.526.485.410]; Cardiovascular Diseases [C14]; Hypertension [C14.907.489]; Hyperlipidemias [C18.452.584.500.500]; Dyslipidemias [C18.452.584.500]; Obesity [C18.654.726.500]; Diabetes Mellitus [C18.452.394.750]; Tobacco Use Disorder [C25.775.912]; Overweight [C23.888.144.699]
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Hyperlipidemias; Dyslipidemias; Obesity; Diabetes Mellitus; Tobacco Use Disorder; Overweight

STUDY DESIGN:
Intervention Model Description: The implementation of the CV Toolkit will be evaluated using a non-randomized stepped wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active implementation of the CV Toolkit (Experimental): The investigators will use a non-randomized stepped wedge design to evaluate the implementation in four VA Women's Practice Based Research Network sites. In this design, the intervention is "turned on" when a primary care provider at the site first engages in the Cardiovascular (CV) Toolkit (i.e. uses a CV screening template which maps to the patient CV self-screener). This design relies on sequential roll-out to participating sites over time, while using other sites as controls until they begin implementation. - The non-randomized design explicitly considers the timing of implementation spread and addresses the statistical issues introduced by lack of randomization in implementation starts and processes. The investigators will analytically compensate for the design by collecting patient-, provider-, and site-level data that may be associated with timing of the adoption of each intervention.
  Interventions: Behavioral: CV Toolkit Components

INTERVENTIONS:
Behavioral: CV Toolkit Components — * Patient completes a CV self screener.
  * Patient discusses CV risks factors with primary care providers and CV risks are documented and discussed for action steps and referrals.
  * Patient will be recommended to attend a gender tailored facilitated workgroup - Gateways to Healthy Living to make specific SMART goals and commit to patient preferred services or program

SUMMARY:
Cardiovascular (CV) disease is the number one cause of death in American women, and all adult women are potentially at risk for CV disease. There are clear gender differences in the control of CV risk factors such as lipids, blood pressure, and intermediate diabetes outcomes nationally and within the VA, with women Veterans often at higher CV risk than their male counterparts. The combination of disparities and gender-specific CV risk factors suggest an urgent need for CV risk factor management in women Veterans. As one project in the Enhancing Mental and Physical health of Women through Engagement and Retention (EMPOWER) QUERI, the objectives of "Facilitating Cardiovascular Risk Screening and Risk Reduction in Women Veterans" are to implement and evaluate a CV risk reduction toolkit (CV toolkit) designed to increase identification of CV risk among Women Veterans, enhance patient/provider communication about their risk, and increase Women Veterans' engagement and retention in relevant health services including referrals to key health programs (e.g., MOVE!, dieticians, health coaches, and CV specialists as needed). The initial CV Toolkit includes four components: (1) Patient education/activation tools including educational materials and a patient CV self-screener to help make CV risk discussion a priority for women before they enter the exam room; (2) A CV risk assessment computerized template to systematically capture CV disease risk factor history and data from the medical record and then facilitate referrals to Gateway to Healthy Living program and other CV risk reduction services/programs; (3) Provider information and education programs as well as referral tools to internal services; and (4) The Gateway to Healthy Living, a facilitated goal-setting group tailored for women Veterans. The goal is to implement the CV Toolkit at four VA facilities with comprehensive women's health clinics. The implementation of the CV Toolkit will be evaluated using a non-randomized stepped wedge design and will apply the evidence-based Replicating Effective Programs (REP) implementation strategy. For the nonrandomized stepped wedge design, each phase represents when one site moved from inactive to active implementation. It was pre-specified for the non-randomized design to evaluate the outcomes as the odds ratio of active intervention versus inactive for the overall study period and not by individual site/phase. This is a function of the use of the non-randomized design. Since the order of sites being introduced into the active intervention is not random, probabilistically the individual site results are not as meaningful here as they would be in a randomized stepped wedge design. Also, mixed methods implementation evaluations will focus on investigating primary implementation outcomes of adoption, acceptability, feasibility, and reach. Multilevel stakeholder engagement will be prioritized. Program-wide organizational-, provider-, and patient-level measures and tools will be utilized to enhance synergy, productivity, impact and facilitate spread.

DETAILED DESCRIPTION:
Background: Women Veterans are the fastest growing segment of Veterans Health Administration (VHA) users. This dramatic growth has created challenges for VHA. Gender disparities persist in cardiovascular (CV) and diabetes risk factor control, and rates of depression, anxiety, and mental health comorbidity are disproportionately high among women Veterans. Furthermore, a high rate of women Veterans' attrition from VA care, along with organizational barriers to care, substantiate that organizational changes are needed in order to engage and retain women Veteran VHA users in evidence-based, patient-centered care.

Objectives: The Enhancing Mental and Physical health of Women through Engagement and Retention (EMPOWER) QUERI addresses VHA Blueprint for Excellence Strategy 6, by advancing "personalized, proactive, patient-centered" care models, and Transformational Strategy 7.2.g by implementation of innovative care models in women Veterans' health care. The EMPOWER QUERI Program is designed to improve women Veterans' engagement and retention in evidence-based care for three high priority health conditions, i.e., prediabetes, cardiovascular, and mental health. To achieve this impact goal, we propose a cohesive portfolio of projects with the following aims: (1) To use an evidence-based implementation strategy that emphasizes local tailoring of care models, multilevel stakeholder engagement, and systematic evaluation of complex implementation processes in order to enrich organizational capacity for innovations in women Veterans' VHA health care; (2) To implement personalized, proactive, patient-centered innovations in VHA women's health that are acceptable, feasible, satisfactory, relevant, and effective for both providers and patients, thereby encouraging women Veterans' engagement and retention and sustainability of the innovations; and, (3) To generate implementation "playbooks" for our partners that are scalable and serve as guidance for future implementation of a broader array of evidence-based women's health programs and policy.

Methods: Three projects will be conducted by an experienced multidisciplinary team. "Tailoring VA's Diabetes Prevention Program to Women Veterans' Needs" is a one-year QI project to be conducted in VA Greater Los Angeles women's health clinics. Women Veterans with prediabetes will select an in-person, peer-led or online gender-specific, evidence-based diabetes prevention program to address their risk behaviors and health conditions. "Facilitating Cardiovascular Risk Screening and Risk Reduction in Women Veterans" will increase identification of CV risk among women Veterans, enhance patient/provider communication and shared decision-making about CV risk, and provide a supportive, coordinated health coaching intervention to facilitate women Veterans' engagement and retention in appropriate health services. "Implementation of Tailored Collaborative Care for Women Veterans" will evaluate implementation of an evidence-based collaborative care model tailored to enhance provider- and system-level capabilities to address women Veterans' anxiety and depression treatment needs, thereby improving organizational primary care-mental health integration (PC-MHI) effectiveness and women Veterans' engagement and retention in PC-MHI. Both implementation research studies will use a non-randomized stepped wedge design and will apply the evidence-based Replicating Effective Programs (REP) implementation strategy. For the nonrandomized stepped wedge design, each phase represents when one site moved from inactive to active implementation. It was pre-specified for the non-randomized design to evaluate the outcomes as the odds ratio of active intervention versus inactive for the overall study period and not by individual site/phase. This is a function of the use of the non-randomized design. Since the order of sites being introduced into the active intervention is not random, probabilistically the individual site results are not as meaningful here as they would be in a randomized stepped wedge design. Mixed methods implementation evaluations will focus on investigating primary implementation outcomes of adoption, acceptability, feasibility, and reach. Multilevel stakeholder engagement will be prioritized. Program-wide organizational-, provider-, and patient-level measures and tools will be utilized to enhance synergy, productivity, and impact. The original protocol proposes the administration of a follow-up survey that includes four secondary outcome measures (PROMIS Global Health; Patient Satisfaction; Overall Anxiety Severity and Impairment Scale (OASIS); and Depression Screen (PHQ-4)). However, the follow-up survey was not administered (data not collected) due to patient burden and COVID-19. As a coherent program of women's health implementation research and quality improvement, the proposed EMPOWER QUERI will constitute a major milestone in achieving BPE strategies and realizing women Veterans' engagement and, ultimately, empowerment in our VHA system.

ELIGIBILITY:
Inclusion Criteria:

* For Patient Activities: Women VA patients with any cardiovascular risk factors
* For Key Stakeholder Activities: VA staff affiliated with the Women's Health Clinic

Exclusion Criteria:

* For Patient Activities: Men & Patients with cognitive impairment precluding informed consent
* For Key Stakeholder Activities: non- VA staff

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6009 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bevanne A Bean-Mayberry, MD MHS, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Melissa M Farmer Coste, PhD MS, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (4):
- United States (4):
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farmer MM, Hamilton AB, Finley EP, Lee ML, Chanfreau C, Than C, Brunner J, Schweizer CA, Moin T, Bean-Mayberry B. Implementation of a cardiovascular toolkit in primary care increased women Veterans' engagement in behavior change programs: results from a non-randomized stepped wedge trial. BMC Prim Care. 2026 Jan 8. doi: 10.1186/s12875-025-03158-5. Online ahead of print. PMID 41507799
- [Derived] Farmer MM, Hamilton AB, Finley EP, Lee M, Chanfreau C, Than C, Brunner J, Schweizer CA, Huynh AK, Moin T, Bean-Mayberry B. Implementation of a cardiovascular toolkit in primary care increased women Veterans' engagement in behavior change programs: results from a non-randomized stepped wedge trial. Res Sq [Preprint]. 2024 Nov 26:rs.3.rs-5347756. doi: 10.21203/rs.3.rs-5347756/v1. PMID 39649163
- [Derived] Clair KS, Bean-Mayberry B, Schweizer CA, Chanfreau C, Jackson L, Than CT, Finley EP, Hamilton A, Farmer MM. Factors Associated with Delayed Care Among Women Veterans Actively Engaged in Primary Care. J Womens Health (Larchmt). 2024 May;33(5):604-612. doi: 10.1089/jwh.2023.0227. Epub 2024 Feb 21. PMID 38386795
- [Derived] Finley EP, Huynh AK, Farmer MM, Bean-Mayberry B, Moin T, Oishi SM, Moreau JL, Dyer KE, Lanham HJ, Leykum L, Hamilton AB. Periodic reflections: a method of guided discussions for documenting implementation phenomena. BMC Med Res Methodol. 2018 Nov 27;18(1):153. doi: 10.1186/s12874-018-0610-y. PMID 30482159
- [Derived] Hamilton AB, Farmer MM, Moin T, Finley EP, Lang AJ, Oishi SM, Huynh AK, Zuchowski J, Haskell SG, Bean-Mayberry B. Enhancing Mental and Physical Health of Women through Engagement and Retention (EMPOWER): a protocol for a program of research. Implement Sci. 2017 Nov 7;12(1):127. doi: 10.1186/s13012-017-0658-9. PMID 29116022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All women with at least one primary care visit at one of the five participating VA clinic sites during the study period (December 2016 - March 2020).
Pre-assignment Details: Non-randomized stepped wedge trial; All women with at least one primary care visit at one of the five participating VA clinic sites during the study period were eligible to receive components of the CV Toolkit when the toolkit was active. Note: one more site implemented the toolkit than the originally proposed four sites.
Units Other Than Participants: Sites
Groups:
- Active Implementation of the CV Toolkit: All women with at least one primary care visit at one of the five participating VA clinic sites during the study period were eligible to receive components of the CV Toolkit when the toolkit was active at their site.
Period: Non-randomized Stepped Wedge Baseline
Arm/Group | Active Implementation of the CV Toolkit
Started | 6009; 5 Sites (CV Template must be completed during time period CV Toolkit is active at the site. Each site had a separate time interval for when the CV Toolkit was active.)
Intervention (Non-active implementation period (control): no sites were actively implementing the CV Toolkit.) | 0; 0 Sites
Control | 6009; 5 Sites
Completed | 6009; 5 Sites
Not Completed | 0; 0 Sites
Period: Trial Step One
Arm/Group | Active Implementation of the CV Toolkit
Started | 6009; 5 Sites
Intervention (First site began active implementation of the CV Toolkit.) | 1461; 1 Sites
Control | 4548; 4 Sites
Completed | 6009; 5 Sites
Not Completed | 0; 0 Sites
Period: Trial Step Two
Arm/Group | Active Implementation of the CV Toolkit
Started | 6009; 5 Sites
Intervention (Second site began active implementation of the CV Toolkit.) | 2704; 2 Sites
Control | 3305; 3 Sites
Completed | 6009; 5 Sites
Not Completed | 0; 0 Sites
Period: Trial Step Three
Arm/Group | Active Implementation of the CV Toolkit
Started | 6009; 5 Sites
Intervention (Third site began active implementation of the CV Toolkit.) | 4909; 3 Sites
Control | 1100; 2 Sites
Completed | 6009; 5 Sites
Not Completed | 0; 0 Sites
Period: Trial Step Four
Arm/Group | Active Implementation of the CV Toolkit
Started | 6009; 5 Sites
Intervention (Fourth site began active implementation of the CV Toolkit.) | 5539; 4 Sites
Control | 470; 1 Sites
Completed | 6009; 5 Sites
Not Completed | 0; 0 Sites
Period: Trial Step Five
Arm/Group | Active Implementation of the CV Toolkit
Started | 6009; 5 Sites
Intervention (Fifth (and final) site began active implementation of the CV Toolkit.) | 6009; 5 Sites
Control | 0; 0 Sites
Completed | 6009; 5 Sites
Not Completed | 0; 0 Sites

BASELINE CHARACTERISTICS:
Population: For the non-randomized stepped wedge analysis, the total population of 6,009 was stratified by age (65+ and less than age 65)
Groups:
- Active Implementation of the CV Toolkit: Women with at least one primary care visit at one of the five participating VA clinic sites during the study period were eligible to receive components of the CV Toolkit when the toolkit was active at their site.
Arm/Group | Active Implementation of the CV Toolkit
Number analyzed (Participants) | 6009
Age, Categorical [Count of Participants; unit: Participants] — Population: For the non-randomized stepped wedge analysis, the total population of 6,009 was stratified by age (65+ and less than age 65)
  Participants
    Stratification: Women Age 65 and Older: number analyzed (Participants) | 618
    Stratification: Women Age 65 and Older: <=18 years | 0
    Stratification: Women Age 65 and Older: Between 18 and 65 years | 0
    Stratification: Women Age 65 and Older: >=65 years | 618
    Stratification: Women Less Than Age 65: number analyzed (Participants) | 5391
    Stratification: Women Less Than Age 65: <=18 years | 0
    Stratification: Women Less Than Age 65: Between 18 and 65 years | 5391
    Stratification: Women Less Than Age 65: >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — All persons identifying as women Population: For the non-randomized stepped wedge analysis, the total population of 6,009 was stratified by age (65+ and less than age 65)
  Participants
    Stratification: Women Age 65 and Older: number analyzed (Participants) | 618
    Stratification: Women Age 65 and Older | 618
    Stratification: Women Less Than Age 65: number analyzed (Participants) | 5391
    Stratification: Women Less Than Age 65 | 5391
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: For the non-randomized stepped wedge analysis, the total population of 6,009 was stratified by age (65+ and less than age 65)
  Participants
    Stratification: Women Age 65 and Older: number analyzed (Participants) | 618
    Stratification: Women Age 65 and Older: Hispanic or Latino | 43
    Stratification: Women Age 65 and Older: Not Hispanic or Latino | 549
    Stratification: Women Age 65 and Older: Unknown or Not Reported | 26
    Stratification: Women Less Than Age 65: number analyzed (Participants) | 5391
    Stratification: Women Less Than Age 65: Hispanic or Latino | 968
    Stratification: Women Less Than Age 65: Not Hispanic or Latino | 4193
    Stratification: Women Less Than Age 65: Unknown or Not Reported | 230
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Due to small numbers, American Indian, Alaska Native, Asian, Native Hawaiian, or Other Pacific Islander were collapsed into one group here to protect confidentiality. Population: For the non-randomized stepped wedge analysis, the total population of 6,009 was stratified by age (65+ and less than age 65)
  Participants
    Race (Stratification: Women Age 65 and Older): number analyzed (Participants) | 618
    Race (Stratification: Women Age 65 and Older): American Indian, Alaska Native, Asian, Native Hawaiian, or Other Pacific Islander | 21
    Race (Stratification: Women Age 65 and Older): Black or African American | 162
    Race (Stratification: Women Age 65 and Older): White | 371
    Race (Stratification: Women Age 65 and Older): Unknown or Not Reported | 64
    Race (Stratification: Women Less Than Age 65): number analyzed (Participants) | 5391
    Race (Stratification: Women Less Than Age 65): American Indian, Alaska Native, Asian, Native Hawaiian, or Other Pacific Islander | 355
    Race (Stratification: Women Less Than Age 65): Black or African American | 1743
    Race (Stratification: Women Less Than Age 65): White | 2583
    Race (Stratification: Women Less Than Age 65): Unknown or Not Reported | 710
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Northeast | 1243
  United States: West | 3666
  United States: South | 1100
  United States: Midwest | 0
Clinic Type [Count of Participants; unit: Participants] — Population: For the non-randomized stepped wedge analysis, the total population of 6,009 was stratified by age (65+ and less than age 65)
  Participants
    Stratification: Women Age 65 and Older: number analyzed (Participants) | 618
    Stratification: Women Age 65 and Older: Women's Clinic | 469
    Stratification: Women Age 65 and Older: Primary Care | 149
    Stratification: Women Less Than Age 65: number analyzed (Participants) | 5391
    Stratification: Women Less Than Age 65: Women's Clinic | 4440
    Stratification: Women Less Than Age 65: Primary Care | 951

OUTCOME MEASURES:

1. Primary Outcome: New Participation in MOVE! (Among Women Aged 65 and Older)
Description: The study utilized a non-randomized stepped wedge design, and in this design, there are two arms: the not-active CV Toolkit arm and the active ("turned on") CV Toolkit arm. All five sites were in both arms at some point in the study period. The determination of when a study was in a particular arm was determined using the non-randomized step wedge design. In this design, all sites begin in the not-active arm and then cross-over to the active arm at a time when they are organized to do so (not a random event). In the non-randomized stepped wedge design (which is very similar to the crossover clinical trial) results are not analyzed separately by arm as is done for standard randomized controlled trials. The analysis also considered stratification of the women by age (< and ≥ 65 years of age). The main outcomes examined participation in MOVE! and HPDP and/or CIH services for each age strata.
Time Frame: 46 months
Population: Comparing participation in MOVE at all 5 sites when CV Toolkit was active (turned one) versus not active (model stratified to include women aged 65 and older only) It was pre-specified in the non-randomized design analysis plan to evaluate the primary outcome measures as the odds ratio between the active and inactive intervention for the overall study period and not by individual site/phase.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Active Implementation of the CV Toolkit
Number analyzed (Participants) | 618
Odds Ratio | 1.09 [1.030 to 1.152]
Statistical Analysis 1: Comparison: Active Implementation of the CV Toolkit; Test type: Superiority; p = .003, Non-linear model with Logit; Non-linear model with Logit Link Function with Robust Standard Errors; Odds Ratio (OR) = 1.09, 95% CI 2-sided [1.030 to 1.152]

2. Primary Outcome: New Participation in MOVE! (Among Women Less Than 65 Years Old)
Description: as for outcome 1
Time Frame: 46 months
Population: Comparing participation in MOVE at all 5 sites when CV Toolkit was active (turned one) versus not active (model stratified to include women less than age 65 only) It was pre-specified in the non-randomized design analysis plan to evaluate the primary outcome measures as the odds ratio between the active and inactive intervention for the overall study period and not by individual site/phase.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Active Implementation of the CV Toolkit
Number analyzed (Participants) | 5391
Odds Ratio | 1.00 [0.976 to 1.022]
Statistical Analysis 1: Comparison: Active Implementation of the CV Toolkit; Test type: Superiority; p = 0.91, Non-linear model with Logit; Non-linear model with Logit Link Function with Robust Standard Errors; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.976 to 1.022]

3. Primary Outcome: Participation in HPDP/CIH Programs (Among Women Aged 65 and Older)
Description: as for outcome 1
Time Frame: 46 months
Population: Comparing participation in HPDP and CIH services at all 5 sites when CV Toolkit was active (turned one) versus not active (model stratified to include women aged 65 and older only) It was pre-specified in the non-randomized design analysis plan to evaluate the primary outcome measures as the odds ratio between the active and inactive intervention for the overall study period and not by individual site/phase.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Active Implementation of the CV Toolkit
Number analyzed (Participants) | 618
Odds Ratio | 1.06 [0.959 to 1.165]
Statistical Analysis 1: Comparison: Active Implementation of the CV Toolkit; Test type: Superiority; p = .265, Non-linear model with Logit; Non-linear model with Logit Link Function with Robust Standard Errors; Odds Ratio (OR) = 1.06, 95% CI 2-sided [.959 to 1.165]

4. Primary Outcome: Participation in HPDP/CIH Programs (Among Women Less Than 65 Years Old)
Description: as for outcome 1
Time Frame: 46 months
Population: Comparing participation in HPDP and CIH services at all 5 sites when CV Toolkit was active (turned one) versus not active (model stratified to include women less than age 65 only) It was pre-specified in the non-randomized design analysis plan to evaluate the primary outcome measures as the odds ratio between the active and inactive intervention for the overall study period and not by individual site/phase.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Odds Ratio
Arm/Group | Active Implementation of the CV Toolkit
Number analyzed (Participants) | 5391
Odds Ratio | 1.01 [1.002 to 1.022]
Statistical Analysis 1: Comparison: Active Implementation of the CV Toolkit; Test type: Superiority; p = 0.015, Non-linear model with Logit; Non-linear model with Logit Link Function with Robust Standard Errors; Odds Ratio (OR) = 1.01, 95% CI 2-sided [1.002 to 1.022]

ADVERSE EVENTS:
Description: Given the nature of this study, adverse advents were not monitored. CV Toolkit was a clinic based intervention and was deemed low/minimal risk by the IRB.
Groups:
- Active Implementation of the CV Toolkit: All women who had a VA visit to a primary care or women's clinic at any of the 5 VA sites while the CV toolkit was being implemented across sites
Arm/Group | Active Implementation of the CV Toolkit
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Additional implementation outcomes (e.g. provider level) were assessed using qualitative methods and will be reported elsewhere (e.g. final report, manuscripts).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT02991534/Prot_SAP_000.pdf